CLINICAL TRIAL: NCT06050733
Title: The Gut Microbiome and Immunotherapy Response in Solid Cancers
Status: Recruiting | Type: Observational
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Other Study IDs: 23-0028
Record Dates: First submitted 2023-09-15; First posted 2023-09-22 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Solid cancer patients with disease progression: 8 patients with a diagnosis of solid cancer undergoing standard of care treatment, with a PD-1 or PD-L1 inhibitor, with disease progression as defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 guidelines.
- Solid cancer patients with stable or experience shrinkage in tumor size: 8 patients with a diagnosis of solid cancer undergoing standard of care treatment, with a PD-1 or PD-L1 inhibitor, with tumor size stable or shrinkage, as defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 guidelines.

SUMMARY:
The aim of this study is characterize the gastrointestinal microbiomes of patient with solid cancer undergoing standard of care treatment with programmed cell death protein 1 (PD-1) /programmed cell death ligand (PD-L1) blockade.

DETAILED DESCRIPTION:
Frontline treatment for solid cancers such as renal cell carcinoma includes immunotherapies such as immune checkpoint inhibitor (ICI) therapy. Despite an increase in overall survival in cancer patients undergoing ICI therapy, many patients' tumors are unresponsive or eventually progress. Recent studies indicate that the gut microbiome composition is associated with clinical response to ICI treatment. Following the success of preclinical research, two recent studies investigated the efficacy of fecal microbiota transplant (FMT) from cancer patients responsive to programmed cell-death protein 1 (PD-1) blockade, a type of ICI treatment, to patients nonresponsive to treatment. Notably, 30-40% of the FMT recipients in these studies subsequently responded to anti-PD-1 therapy. However, the effectiveness of FMT may vary among donors, there is no clear agreement on the ideal FMT composition, and FMT carries the risk of transmitting infection. An alternative to FMT is identification of specific efficacious commensals for supplementation. While the specific commensals enriched in cancer patients with more favorable outcomes vary from study to study, several are commonly reported, including Akkermansia muciniphila, Bacteroides spp., Bifidobacterium spp., Ruminococcaceae spp., and Faecalibacterium spp.

Cancer-related fatigue is experienced by nearly all patients during treatment, and cancer-related cognitive impairment (CRCI), which is a decrease in neurocognitive functioning that can be caused by cancer or its treatment, is present in up to ¾ of patients during treatment. Fatigue and CRCI have both been linked to the composition of the gut microbiome in cancer patients.

Specific Aims

Specific Aim 1: Characterize the gut microbiome of solid cancer patients that have had disease progression during standard-of-care treatment with PD-1 or programmed cell death ligand 1 (PD-L1) blockade and compare to solid cancer patients that were stable or experienced tumor shrinkage during standard-of-care treatment with PD-1/PD-L1 blockade.

Specific Aim 2: Assess neuropsychological measures of cognition and fatigue in solid cancer patients undergoing standard-of-care treatment with PD-1/PD-L1 blockade and determine associations with composition of the gut microbiome.

ELIGIBILITY:
Inclusion Criteria:

1. Current diagnosis of malignant solid cancer that is nonresectable or metastatic.
2. Ages 35 to 75 years.
3. Treatment with immunotherapy, specifically programmed cell death protein 1 (PD-1) or programmed cell death ligand 1 (PD-L1) inhibitor, for at least 3 months but less than 24 months (except for previously responsive subjects re-enrolling as non-responsive patients).
4. Measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 guidelines.
5. Participant is willing and able to give informed consent for participation in the study

Exclusion Criteria:

1. Significant heart, liver, blood or respiratory disease.
2. Current diagnosis of HIV, Hepatitis B or Hepatitis C.
3. History of heart disease.
4. Uncontrolled diabetes mellitus.
5. Subjects with a history of inflammatory bowel disease, Celiac disease or active diverticular disease.
6. Females who are pregnant or lactating.
7. Treatment with chemotherapy within the past 2 years.
8. Treatment with kinase inhibitors within the past 3 months.
9. Previous radiation therapy for brain metastases.
10. Other medical condition or medication administration deemed exclusionary by the study investigators.

Ages: 35 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients from cancer clinic
Sampling Method: Non-Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2023-06-30 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Characterization of fecal microbiome using molecular methods | baseline
  Characterization of the fecal microbiome using a commercially available sampling kit and our lab's patented array for PCR.

SECONDARY OUTCOMES:
Cognitive Function as measured by Montreal Cognitive Assessment | baseline
  The Montreal Cognitive Assessment (MoCA) will be used to assess cognition.
  The Montreal Cognitive Assessment (MoCA) is a rapid assessment of cognition. The MoCA consists of 9 questions with the following subcategories: visuospatial/executive, naming, memory, language, abstraction, delayed recall and orientation. The MoCA has been used extensively to detect cognitive impairment in many conditions, including head trauma. Version 7.1 will be used. Scores range from 0 to 30, higher score being a better outcome.
Fatigue as measured by the Multidimensional Fatigue Symptom Inventory | baseline
  Multidimensional Fatigue Symptom Inventory Short Form (MFSI-SF) from the Moffitt Cancer Center, University of South Florida The MFSI-SF is a 30 question assessment designed to assess the principal manifestations of fatigue.
  There 5 subscales used to calculate a total score. The subscales are: General Fatigue, Physical Fatigue, Emotional Fatigue, Mental Fatigue, and Vigor (an estimate of the patient's energy level). The total score is calculated with the equation: (general + physical + emotional + mental) - vigor = total score.
  The range of the total score is -24 to 96, with the higher the number meaning more fatigue.
Fatigue and Cognition as measured by the Fatigue and Altered Cognition Scale | baseline
  The Fatigue and Altered Cognition Scale (FACS) is a joint project from University of Texas Medical Branch and Texas A&M University. The FACS is a 20 question assessment designed to access perceived fatigue and cognition.
  There are 2 subscales used to calculate a total score. The subscales are: Fatigue and Altered Cognition. The total score is calculated by adding the subscales together. The range of the total score is 0-100, with a higher score indicating more fatigue and altered cognition.
Gastrointestinal Health measured by the Gastrointestinal Symptom Rating Scale | baseline
  The Gastrointestinal Symptom Rating Scale (GSRS) is a specific 15-item questionnaire. Subjects are asked to numerically score their subjective symptoms on a scale of 1-7 (1 = no discomfort at all; 7 = very severe discomfort) . The sum of the scores for all 15 items is regarded as the GSRS total score. Total scores range from 15 (best outcome) to 105 (worst outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Melinda Sheffield-Moore, PhD, Principal Investigator — University of Texas
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No